CLINICAL TRIAL: NCT06248307
Title: Evaluación Del Efecto de la Ingesta de Una Barrita Con Alto Contenido de proteína Sobre el Peso y la Salud Osteoarticular
Brief Title: Evaluation of Protein Bars on Weight Management and Osteoarthicular Health
Acronym: COLARTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Viscofan (Industry)
Responsible Party: Principal Investigator, Santiago Navas, Principal Investigator, University of Navarra
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COLARTIC
Record Dates: First submitted 2024-01-30; First posted 2024-02-08 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Overweight and Obesity; Articular Disease
Keywords: Nutritional intervention
MeSH Terms: conditions — Overweight; Obesity; Joint Diseases

STUDY DESIGN:
Intervention Model Description: 2 parallel groups, double-blind, randomized intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Barrita experimental (Experimental): Two bars to be consumed before lunch and before dinner
  Interventions: Dietary Supplement: Barrita experimental
- Barrita placebo (Placebo Comparator): Two bars to be consumed before lunch and before dinner
  Interventions: Dietary Supplement: Barrita Placebo

INTERVENTIONS:
Dietary Supplement: Barrita experimental — Nutritional advice, as well as administration of protein bars.
  Arms: Barrita experimental
Dietary Supplement: Barrita Placebo — Nutritional advice, as well as administration of placebo bars.
  Arms: Barrita placebo

SUMMARY:
The goal of this intervention study is to evaluate the efficacy in subjects with overweight or obesity of protein bars consumption. The main questions it aims to answer are:

* Does the regular consumption of these protein bars help to loose weight?
* Does the regular consumption of these protein bars help to improve the osteoarticular health? Participants will be asked to follow the indications of consumption of the bars togather with healthy nutritional advice during 16 weeks.

Researchers will compare exparimental Versus placebo groups to see if weight is lost in similar or different ways.

DETAILED DESCRIPTION:
The intervention is designed to evaluate the efficacy of the consumption of a protein bar vs placebo on weight control and osteoarticular health.

For this purpose, a total of 102 subjects will be randomised to either the experimental group or the placebo group, the only stratification performed will be acording to sex.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 37.5 kg/m2
* Normal physical examination and vital signs according to clinical examiners.
* Chronic pharmacological treatment is permitted if dosage is stable within at least three months prior the start of the intervention.

Exclusion Criteria:

* Any funcitonal or structural impairment in digestive system (hitus hernia, ulcers, inflammatory bowel disease, etc.)
* Excessive alcohol consumption (> 14 units/week in women and > 20 units per week in men)
* Bariatric surgery or similar
* Arthritis, hepatic diseases, cancer.
* Alergy to any component of the products
* Subjects presenting any cognitive or psichiatric impairment, that may impel them to follow the protocol.
* Subjects following any weight loss program

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Ponderal evolution | 16 weeks
  Change in body weight between baseline and end of intervention
Change in fat mass | 16 weeks
  Body composition . Change in fat mass between baseline and end of intervention
Change in fat-free mass | 16 weeks
  Body composition . Change in fat-free mass between baseline and end of intervention

SECONDARY OUTCOMES:
Osteoarticular changes | 16 weeks
  Measure the knee articular range between baseline and end of intervention
Plasma P2P and CTX-II levels | 16 weeks
  Evaluate changes in markers between baseline and end of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigacion en Nutricion. Universidad de Navarra, Pamplona, Navarre, Spain